CLINICAL TRIAL: NCT01526408
Title: Treatment of Hearing Fluctuation in Unilateral Meniere's Disease: A Randomized, Placebo-controlled Clinical Trial of Famciclovir
Brief Title: Famvir for Treatment of Hearing in Unilateral Meniere's Disease
Acronym: Famvir
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: HRI no longer conducting research.
Sponsor: House Research Institute (Other)
Collaborators: House Clinic, Inc. (Industry)
Responsible Party: Principal Investigator, M. Jennifer Derebery, Principal Investigator, House Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRI-003; Meniere's Disease (Other: House Research Institute)
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Meniere's Disease
Keywords: Meniere's Disease; Vertigo; Hearing loss; Tinnitus; Anti-viral; Famciclovir
MeSH Terms: conditions — Meniere Disease; Vertigo; Hearing Loss; Tinnitus | interventions — Famciclovir

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Arm (Placebo Comparator): Treatment with 3 months of placebo
  Interventions: Drug: Placebo
- Active Arm (Active Comparator): Treatment with 3 months of active drug
  Interventions: Drug: Famciclovir

INTERVENTIONS:
Drug: Famciclovir — Patients will be instructed to take 6 250mg pills orally for the first 7 days (Week 1: 2 pills every 8 hours or three times per day) at home. Patients will take a maintenance dose of one 250 mg pill twice a day for 77 days (11 weeks, total 3 months on drug).
  Other Names: Famvir
  Arms: Active Arm
Drug: Placebo — Patients will be instructed to take 6 250mg pills orally for the first 7 days (Week 1: 2 pills every 8 hours or three times per day) at home. Patients will take a maintenance dose of one 250 mg pill twice a day for 77 days (11 weeks, total 3 months).
  Arms: Placebo Arm

SUMMARY:
The specific aim of this study is to determine the efficacy of treatment with famciclovir in unilateral Meniere's Disease patients, specifically whether hearing can be improved. The investigators will determine the percentage of unilateral Meniere's Disease patients experiencing an absence of hearing fluctuation after 3 months of treatment with famciclovir as compared to the placebo arm.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral Meniere's Disease
* 2 vertigo episodes of at least 20 minutes
* Fluctuating hearing by subjective history and/or audiometric documentation. Audiometric documentation is defined as affected ear pure-tone average change from an audiogram at Time 1 to Time 2 (less than one year apart) of greater than 15 dB.
* Less than 45 dB 4-frequency pure-tone average in the affected ear
* Tinnitus and/or aural fullness
* Willing to undergo the clinical trial procedures
* Signed informed consent

Exclusion Criteria:

* Acute or chronic middle ear disease in either ear
* Only hearing ear
* 4-frequency pure-tone average > 45 dB in either ear
* Known allergy to famciclovir or any of the ingredients in the formulation
* Taking oral steroids or receiving IT steroids at time of enrollment. If the subject has been on oral steroids/IT steroids, 3 months must elapse from last dose to start of treatment in the study
* Must not have had previous inner ear surgery
* History of immunodeficiency diseases such as HIV
* History of renal insufficiency or other kidney diseases
* A female of child-bearing potential who is pregnant
* History of noncompliance to medical regimens
* Unwilling to or unable to comply with the protocol, including scheduling study evaluations

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-12; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Derebery, MD, Principal Investigator — House Research Institute

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Arm | Active Arm
Started | 0 (early termination of study and sponsor organization closed) | 0 (early termination of study and sponsor organization closed)
Completed | 0 (early termination of study and sponsor organization closed) | 0 (early termination of study and sponsor organization closed)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: early termination of study and sponsor organization closed
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Arm | Active Arm | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Pure-tone Threshold Change
Description: Change in hearing from baseline to after 3 months of treatment
Time Frame: 3 months
Population: early termination of study and sponsor organization closed
Arm/Group | Placebo Arm | Active Arm
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Tinnitus and/or Dizziness Handicap Change
Description: Change in tinnitus and/or dizziness from baseline to after 3 months of treatment
Time Frame: 3 months
Population: early termination of study and sponsor organization closed
Arm/Group | Placebo Arm | Active Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: early termination of study and sponsor organization closed
Description: early termination of study and sponsor organization closed
Arm/Group | Placebo Arm | Active Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes